CLINICAL TRIAL: NCT02942342
Title: Evaluation of Asymptomatic Coronary Atherosclerotic Disease Among People of Kalamazoo County and Neighboring Areas in Michigan, Who Have Risk Factors of Coronary Artery Disease
Brief Title: Evaluation of Asymptomatic Coronary Atherosclerotic Disease Among People of Kalamazoo, MI
Acronym: ESCAPE MI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Borgess Research Institute (Other)
Responsible Party: Principal Investigator, Vishal Gupta, Medical Director, Cardiac Catheterization Laboratory, Borgess Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-2466
Record Dates: First submitted 2016-03-31; First posted 2016-10-24 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Coronary Artery Disease; Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

INTERVENTIONS:
Procedure: Computed Tomography (CT) Scan — CT Scans will be used as a diagnostic tool for asymptomatic CAD.

SUMMARY:
The primary goal of this study is to determine the prevalence of undiagnosed asymptomatic coronary artery disease (CAD) in Kalamazoo and its neighboring areas using Coronary Computed Tomography (CCTA) and Coronary Artery Calcium Score (CACS) to assess if asymptomatic CAD is widespread enough to warrant implementation of CCTA as a routine screening tool. Additionally, this study will use the CCTA results to evaluate several methods of assessing CAD risk in the asymptomatic population including Framingham Risk Score (FRS) and Reynold's Risk Score, Biomarkers (High sensitivity C-Reactive Protein, Fibrinogen, Vertical Auto Profile, oxidized Low Density Lipoprotein (LDL), Apolipoprotein A1 (ApoA1), Apolipoprotein B1 (ApoB1), Vitamin D, Homocysteine) as well as a large panel of genetic markers of atherosclerosis and dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 35 and 55 years of age.
2. Subject receives care in Kalamazoo County and neighboring areas.
3. No known history of coronary artery disease, peripheral vascular disease or stroke.
4. Asymptomatic per shortened World Health Organization (WHO) Rose Angina Questionnaire.
5. Any one of the following sets of clinical risk factors for CAD:

   1. Premature Immediate Family History of CAD (Male <55 years old, Female <65 years old)
   2. Diabetes Mellitus Type 2
   3. Chronic Smoker (currently smoking at least 1 cigarette per month)
   4. Any family history of CAD with Dyslipidemia or hypertension or former smoker
6. Stress test or cardiac catheterization procedure is not clinically indicated for the subject at the time of enrollment.
7. Subject has signed informed consent.

Exclusion Criteria:

1. Subject has known coronary artery disease.
2. Known abnormal stress test where coronary angiography is indicated.
3. Subject is unable to routinely walk at least 20 feet without assistance (e.g., requires a walker or wheelchair to mobilize or has known paralysis).
4. Subject reports they have active systemic or cutaneous infection or inflammation (e.g., septicemia at the time of the procedure).
5. Subject has uncontrolled hypertension (> 180 mmHg systolic and >110mmHg diastolic).
6. Subject presents with hemodynamic instability or is in need of emergent surgery.
7. Known contraindications or known severe reaction to iodinated contrast media.
8. Known contraindications to beta-blockers.
9. Known contraindications to use of sublingual nitroglycerine.
10. Subject has history of chronic kidney disease, with a Glomerular Filtration Rate (GFR) of 45 or below.
11. Subject has known history of Non-Ischemic Cardiomyopathy (NICMP)
12. Subject has a pre-existing severe systemic disease or illness that results in an expected life expectancy of less than 2 years.
13. Subject is currently participating in an investigational drug or another device study that clinically interferes with the current study endpoints.
14. Pregnant or lactating subjects.
15. Known arrhythmias that does not allow electrocardiogram (ECG) triggering, as determined at the time of CT scan. ECG prior to procedure is not indicated.
16. History of a brain tumor; a recent (within the past 6 months) head or brain injury, concussion, epilepsy, or other seizure disorders, severe liver disease, sickle cell anemia, multiple sclerosis, substance abuse, multiple myeloma, pheochromocytoma, or a thyroid disorder.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-03; Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Estimation of the proportion of people in the Kalamazoo, MI, area who have asymptomatic CAD. | 3 years
Compare evidence of atherosclerosis or calcification, as evidenced by CT scan, to associated biomarker values. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Vishal Gupta, MD, MPH, Principal Investigator — Borgess Medical Center
Locations (1):
- Borgess Medical Center, Kalamazoo, Michigan, United States